CLINICAL TRIAL: NCT01142115
Title: Comparative Study of Two Different Urine Catheters.
Brief Title: Test of Discomfort and Malaise of Two Different Urine Catheters in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CP063CC
Record Dates: First submitted 2010-05-04; First posted 2010-06-11 (Estimated); Results first posted 2011-08-09 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monza (Experimental): nonCE marked intermittent catheter
  Interventions: Device: Intermittent catheter CP063CC
- control (Active Comparator): SpeediCath coated catheter
  Interventions: Device: Intermittent catheter CP063CC; Device: SpeediCath

INTERVENTIONS:
Device: Intermittent catheter CP063CC — intermittent catheterisation
  Other Names: Intermittent catheter,
Device: SpeediCath — intermittent catheterisation
  Other Names: Intermittent catheter
  Arms: control

SUMMARY:
The purpose of this study is to evaluate the safety of a new developed catheter in comparison with an catheter on the market. The study is randomised.

DETAILED DESCRIPTION:
Intermittent catheterization is the preferred method for emptying the bladder in patients with spinal cord injury and neurogenic bladder dysfunction.

Coloplast has developed a new intermittent catheter. In this investigation this new test catheter will be compared with SpeediCath by assessing discomfort and pain associated with catheterization of healthy men. The reason for choosing healthy men is that many catheter users do not have full feeling in their urethra and therefore can not assess the discomfort.

Healthy men who are ≥ 18 years and have no signs of urinary tract infection and do not have abnormalities, disease or have had operational interventions in the urinary tract will be included. They are recruited through advertisements on the website www.forsoegsperson.dk.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Male
* signed informed Consent,
* Neg. urine multistix

Exclusion Criteria:

* Abnormalities,
* diseases or surgical procedures performed in the lower urinary-tract

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rikke Otttesen, CTM, Study Director — Coloplast A/S
Locations (1):
- Rigshospitalet, dep. 2112, Copenhagen, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: January-May, 2010, Department of Urology, Rigshospitalet, Denmark
Groups:
- SpeediCath First, Then Monza: Catheterization with SpeediCath catheter on visit 1. Catheterization with Monza catheter on visit 2.
- Monza First, Then SpeediCath: Catheterization with Monza catheter on visit 1. Catheterization with SpeediCath catheter on visit 2.
Period: First Intervention
Arm/Group | SpeediCath First, Then Monza | Monza First, Then SpeediCath
Started | 21 | 20
Completed | 19 | 19
Not Completed | 2 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Adverse Event | 1 | 0
Period: Second Intervention
Arm/Group | SpeediCath First, Then Monza | Monza First, Then SpeediCath
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive SpeediCath first and Monza first
Arm/Group | Entire Study Population
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25.9 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 41
Region of Enrollment [Number; unit: participants]
  Denmark | 41

OUTCOME MEASURES:

1. Primary Outcome: Discomfort Measured on the Visual Analog Scale (VAS)
Description: Outcome measured on a 10 cm Visual Analog Scale ranging from "no discomfort" (0cm) to "worst thinkable discomfort" (10cm).
Time Frame: 10 minutes after each catheterisation at visit 1 and at visit 2 which is 5-25 days after visit 1
Population: Intention to Treat (ITT) population
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Monza: Test product
- SpeediCath: Control Product
Arm/Group | Monza | SpeediCath
Number analyzed (Participants) | 38 | 39
cm | 3.7 (2.2) | 2.6 (1.8)
Statistical Analysis 1: Comparison: Monza vs SpeediCath; Test type: Non-Inferiority or Equivalence — The estimated difference VAS(Monza) minus VAS(SpeediCath)(i.e. the upper confidence limit) shall be less than 1cm to demonstrate non-inferiority; p = 0.0018, Mixed Models Analysis; Mean Difference (Final Values) = 1.052, 95% CI 2-sided [0.412 to 1.692]

2. Secondary Outcome: Irritation During Voiding After Catheterization
Description: After each catheterization subjects were asked if they felt any irritation during voiding with answer option yes or no.
  Yes - they experienced irritation. No - they did not experience irritation.
Time Frame: 10 minutes after each catheterization at visit 1 and at visit 2, which is 5-25 days after visit 1
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Monza | SpeediCath
Number analyzed (Participants) | 38 | 39
Participants
  Answer "Yes" | 21 | 7
  Answer "No" | 17 | 32
Statistical Analysis 1: Comparison: Monza vs SpeediCath; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 5.805, 95% CI 2-sided [2.604 to 12.939]

3. Secondary Outcome: Ease of Use Measured on a 5 Point Scale: Insertion Effort
Description: After each catheterization the nurse who conducted the catheterization answered how the catheter insertion had been.
  There were 5 answer categories: very difficult - difficult - neither easy nor difficult - easy - very easy
Time Frame: 10 minutes after each catheterization at visit 1 and at visit 2, which is 5-25 days after visit 1
Population: ITT
Measure: Number; unit: participants
Arm/Group | Monza | SpeediCath
Number analyzed (Participants) | 38 | 39
participants
  Answer "Very Easy" | 2 | 7
  Answer "Easy" | 16 | 20
  Answer "Neither easy nor difficult" | 13 | 8
  Answer "Difficult" | 6 | 4
  Answer "Very Difficult" | 1 | 0
Statistical Analysis 1: Comparison: Monza vs SpeediCath; Test type: Superiority or Other; p = 0.6160, Proportional odds regression model; Odds Ratio (OR) = 0.822, 95% CI 2-sided [0.382 to 1.767]

4. Secondary Outcome: Ease of Use Measured on a 5 Point Scale: Withdrawal Effort
Description: After each catheterization the nurse who conducted the catheterization answered how the catheter withdrawal had been.
  There were 5 answer categories: very difficult - difficult - neither easy nor difficult - easy - very easy
Time Frame: 10 minutes after each catheterization at visit 1 and at visit 2, which is 5-25 days after visit 1
Population: ITT
Measure: Number; unit: participants
Arm/Group | Monza | SpeediCath
Number analyzed (Participants) | 38 | 39
participants
  Answer "Very Easy" | 28 (0.45) | 28 (0.46)
  Answer "Easy" | 10 | 11
  Answer "Neither easy nor difficult" | 0 | 0
  Answer "Difficult" | 0 | 0
  Answer "Very difficult" | 0 | 0
Statistical Analysis 1: Comparison: Monza vs SpeediCath; Test type: Superiority or Other; p = 0.8014, Proportional odds regression model; Odds Ratio (OR) = 1.117, 95% CI 2-sided [0.472 to 2.646]

5. Secondary Outcome: Visible Blood
Description: Visual blood observed on the catheter or in the urine in connection to catheterization.
  The nurse who conducted the catheterization could answer yes or no as follows:
  Yes = visible blood observed. No = no visible blood observed.
Time Frame: 10 minutes after each catheterization at visit 1 and at visit 2, which is 5-25 days after visit 1
Population: ITT
Measure: Number; unit: participants
Arm/Group | Monza | SpeediCath
Number analyzed (Participants) | 38 | 39
participants
  Visible blood | 3 | 1
  No visible blood | 35 | 38
Statistical Analysis 1: Comparison: Monza vs SpeediCath; Test type: Superiority or Other; p = 0.3085, Regression, Logistic; Odds Ratio (OR) = 3.503, 95% CI 2-sided [0.314 to 39.106]

6. Secondary Outcome: Haematuria
Description: Negative or positive result on a multistix urin analysis.
  Negative haematuria: 10 erythrocytes/microliter or less. Positive haematuria: above 10 erythrocytes/microliter.
Time Frame: 2 hours after catheterisation at visits 1 and 2
Population: ITT
Measure: Number; unit: participants
Arm/Group | Monza | SpeediCath
Number analyzed (Participants) | 38 | 39
participants
  Positive for haematuria | 10 | 9
  Negative for haematuria | 28 | 30
Statistical Analysis 1: Comparison: Monza vs SpeediCath; Test type: Superiority or Other; p = 0.4324, Proportional odds regression model; Odds Ratio (OR) = 1.398, 95% CI 2-sided [0.606 to 3.225]

ADVERSE EVENTS:
Arm/Group | Entire Study Population
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 1/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Entire Study Population (N=41)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) — Not related to the device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other